CLINICAL TRIAL: NCT06506565
Title: A Randomized, Placebo-Controlled, Double-Blind Evaluation of Low-Dose Ketamine Infusion During Burn Wound Care Procedures to Improve Pain Intensity and Reduce Opioid Consumption
Brief Title: Low-Dose Ketamine Infusion During Burn Wound Care
Acronym: IMPROVE
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Tennessee (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 23-09751-FB
Record Dates: First submitted 2024-07-11; First posted 2024-07-17 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Burn; Pain; Dissociation; Opioid
Keywords: ketamine; burn; opioid; analgesia
MeSH Terms: conditions — Burns; Pain; Dissociative Disorders; Agnosia | interventions — Ketamine; Saline Solution

STUDY DESIGN:
Intervention Model Description: Patients will be randomly enrolled by blocks according to age, burn size, and opioid use history. Study treatment will occur for up to 7 days. Assignment will be to placebo or ketamine and all participants and staff will be blinded, except pharmacy. Each patient will receive standard of care fentanyl and midazolam during wound care regardless of study assignment.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All team members and patients are blinded to study treatment, except pharmacy staff.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ketamine (Experimental): Ketamine infusion (0.3 mg/kg/hr) to begin 1 hour before wound care, continuing through and for 1 hour following wound care.
  Interventions: Drug: Ketamine
- Placebo (Placebo Comparator): 0.9% saline to begin 1 hour before wound care, continuing through and for 1 hour following wound care.
  Interventions: Drug: 0.9% NaCl

INTERVENTIONS:
Drug: Ketamine — Infusion during wound care
  Arms: Ketamine
Drug: 0.9% NaCl — Infusion during wound care
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
The current standard of care (SOC) (i.e. fentanyl and midazolam) offers limited efficacy for preventing or relieving pain. Ketamine infusions may provide the benefits of analgesia, minimize adverse events, and reduce opioid use. The purpose of this study is to determine if adding a low dose ketamine infusion during wound care will safely provide pain relief for patients with burn injury.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to burn service with thermal injury

Exclusion Criteria:

* unable/unwilling to consent within 72 hours
* unable to report NRS
* known contraindication to ketamine
* < than 18 years of age
* pregnant
* incarcerated
* TBSA over 50 %

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2024-07-08 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Analgesia | up to 7 days from enrollment
  Numeric Pain Rating Scale (0 - 10, with 0 being absence of pain and 10 being the worst pain imaginable)

CONTACTS AND LOCATIONS:
Locations (1):
- Regional One Health, Memphis, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No